CLINICAL TRIAL: NCT04230928
Title: A Pilot Study Comparing Dietary Approaches to Decrease Hypertension in a Lower Income, African American Population at Risk for Cardiovascular Disease
Brief Title: Giving a Low Carbohydrate Diet to Overcome Hypertension
Acronym: GLOH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 019-268
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hypertension; African Americans; Diet, Carbohydrate-Restricted; Risk Reduction Behavior
Keywords: Hypertension; Low carbohydrate diet; African American race; Cardiovascular disease risk; Weight loss
MeSH Terms: conditions — Hypertension; Risk Reduction Behavior; Weight Loss

STUDY DESIGN:
Intervention Model Description: Prospective randomized 2-group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard GLB Control (Placebo Comparator): Individuals will receive the standard Diabetes Prevention Program-Group Lifestyle Balance (GLB) program as outlined by the American Diabetes Association. This program will be taught at the Baylor Scott & White Health and Wellness Center by trained research staff.
  Interventions: Other: Standard DPP-GLB diet; Behavioral: Standard DPP-GLB program modules
- VLC-GLB Intervention (Experimental): Individuals will receive a version of the DPP-GLB program in which 4 of the 12 modules will teach a very low carbohydrate diet instead of the standard. All other components of the DPP-GLB will follow the standard. This program will be taught at the Baylor Scott & White Health and Wellness Center by trained research staff.
  Interventions: Other: Very low carbohydrate diet; Behavioral: Standard DPP-GLB program modules

INTERVENTIONS:
Other: Very low carbohydrate diet — Participants will learn to follow a very low carbohydrate diet in modified versions of GLB modules 2,3,5 & 10. Participants will learn to track carbohydrate intake
  Arms: VLC-GLB Intervention
Other: Standard DPP-GLB diet — Participants will learn to follow a very low fat, calorie-restricted diet and track fat grams and caloric intake in standard GLB modules 2,3,5, & 10
  Arms: Standard GLB Control
Behavioral: Standard DPP-GLB program modules — Participants will learn standard DPP-GLB modules for other lifestyle modifications for stress, physical activity, etc. in sessions 1,4,6-9, 11-22

SUMMARY:
This study will test the preliminary efficacy of adding a very low carbohydrate dietary intervention to the evidence-based DPP-GLB on blood pressure reductions for lower-income AA men and women in a community-based clinic.

DETAILED DESCRIPTION:
This study will evaluate the effects of consuming a very low carbohydrate (VLC) diet in a sustainable community care setting, in addition to routine medical care, to African American (AA) with pre-hypertension, hypertension (stage 1-3), or cardiovascular disease risk factors. This study will also secondarily assess the feasibility of following a VLC diet in a low-income, AA population.

ELIGIBILITY:
Inclusion Criteria:

* 1) men and women aged ≥ 18 years
* 2) willingness to participate in a 10-month study
* 3) systolic blood pressure > 120 mm/Hg +/- diastolic blood pressure > 80 mm/Hg
* 4) African American race

Exclusion Criteria:

* 1) diagnosed congestive heart failure
* 2) Hypertension stage 4 or higher (e.g., SBP >180 mm/Hg; DBP > 110 mm/Hg)
* 3) received or needing more than 3 anti-hypertensive medications
* 4) pregnant or planning to become pregnant
* 5) receiving or needing a heart transplant
* 6) Using injected long or short-acting insulin for diabetes treatment
* 7) not African American race
* 8) unable to speak and read English with fluency

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Systolic blood pressure | Baseline; 12 weeks; 10 months
  Measure changes in both systolic and diastolic blood pressure using digital sphygmomanometer; NOTE: Only Systolic BP is primary outcome, diastolic change will be a secondary outcome measure
Dietary changes in carbohydrate intake | Baseline; 12 weeks; 10 months
  Assess changes in diet using ASA24 online dietary recall

SECONDARY OUTCOMES:
Changes in Fasting blood glucose | Baseline; 12 weeks; 10 months
  Finger stick measure of blood glucose levels collected after 8-12 hours fasting
Changes in Hemoglobin A1C | Baseline; 12 weeks; 10 months
  Finger stick measure of hemoglobin A1C collected after 8-12 hours fasting
Changes in Cholesterol and lipoproteins | Baseline; 12 weeks; 10 months
  Finger stick measure of blood levels of total cholesterol, HDL, LDL, and triglycerides collected after 8-12 hours fasting
Changes in % Body weight | Baseline; 12 weeks; 10 months
  Change in weight measured in lbs. with digital scale; % change calculated
Changes in Body mass index (BMI) | Baseline; 12 weeks; 10 months
  Change in calculated BMI based upon height (in.) with stadiometer & weight (lbs.) with digital scale
Dietary changes in fat intake | Baseline; 12 weeks; 10 months
  Assess changes in diet using ASA24 online dietary recall
Dietary changes in caloric intake | Baseline; 12 weeks; 10 months
  Assess changes in diet using ASA24 online dietary recall
Changes in Diastolic blood pressure | Baseline; 12 weeks; 10 months
  Measure changes in both systolic and diastolic blood pressure using digital sphygmomanometer; NOTE: Only Systolic BP is primary outcome, diastolic change will be a secondary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Aisha H Montgomery, MD, MPH, Principal Investigator — Baylor Scott and White Health
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies results in publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 6 months of outcome publication

REFERENCES:
- [Background] Gillum RF. Pathophysiology of hypertension in blacks and whites. A review of the basis of racial blood pressure differences. Hypertension. 1979 Sep-Oct;1(5):468-75. doi: 10.1161/01.hyp.1.5.468. PMID 541040
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Lackland DT. Racial differences in hypertension: implications for high blood pressure management. Am J Med Sci. 2014 Aug;348(2):135-8. doi: 10.1097/MAJ.0000000000000308. PMID 24983758
- [Background] Zhang D, Wang G, Zhang P, Fang J, Ayala C. Medical Expenditures Associated With Hypertension in the U.S., 2000-2013. Am J Prev Med. 2017 Dec;53(6S2):S164-S171. doi: 10.1016/j.amepre.2017.05.014. PMID 29153117
- [Background] Howard G, Prineas R, Moy C, Cushman M, Kellum M, Temple E, Graham A, Howard V. Racial and geographic differences in awareness, treatment, and control of hypertension: the REasons for Geographic And Racial Differences in Stroke study. Stroke. 2006 May;37(5):1171-8. doi: 10.1161/01.STR.0000217222.09978.ce. Epub 2006 Mar 23. PMID 16556884
- [Background] Lackland DT, Keil JE. Epidemiology of hypertension in African Americans. Semin Nephrol. 1996 Mar;16(2):63-70. PMID 8668862
- [Background] Kitzman H, Dodgen L, Mamun A, Slater JL, King G, Slater D, King A, Mandapati S, DeHaven M. Community-based participatory research to design a faith-enhanced diabetes prevention program: The Better Me Within randomized trial. Contemp Clin Trials. 2017 Nov;62:77-90. doi: 10.1016/j.cct.2017.08.003. Epub 2017 Aug 12. PMID 28807739
- [Background] Tiwari S, Riazi S, Ecelbarger CA. Insulin's impact on renal sodium transport and blood pressure in health, obesity, and diabetes. Am J Physiol Renal Physiol. 2007 Oct;293(4):F974-84. doi: 10.1152/ajprenal.00149.2007. Epub 2007 Aug 8. PMID 17686957
- [Background] Meckling KA, Gauthier M, Grubb R, Sanford J. Effects of a hypocaloric, low-carbohydrate diet on weight loss, blood lipids, blood pressure, glucose tolerance, and body composition in free-living overweight women. Can J Physiol Pharmacol. 2002 Nov;80(11):1095-105. doi: 10.1139/y02-140. PMID 12489929
- [Background] Rehm CD, Penalvo JL, Afshin A, Mozaffarian D. Dietary Intake Among US Adults, 1999-2012. JAMA. 2016 Jun 21;315(23):2542-53. doi: 10.1001/jama.2016.7491. PMID 27327801
- [Background] Saslow LR, Kim S, Daubenmier JJ, Moskowitz JT, Phinney SD, Goldman V, Murphy EJ, Cox RM, Moran P, Hecht FM. A randomized pilot trial of a moderate carbohydrate diet compared to a very low carbohydrate diet in overweight or obese individuals with type 2 diabetes mellitus or prediabetes. PLoS One. 2014 Apr 9;9(4):e91027. doi: 10.1371/journal.pone.0091027. eCollection 2014. PMID 24717684
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Yancy WS Jr, Westman EC, McDuffie JR, Grambow SC, Jeffreys AS, Bolton J, Chalecki A, Oddone EZ. A randomized trial of a low-carbohydrate diet vs orlistat plus a low-fat diet for weight loss. Arch Intern Med. 2010 Jan 25;170(2):136-45. doi: 10.1001/archinternmed.2009.492. PMID 20101008
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Armstrong C; Joint National Committee. JNC8 guidelines for the management of hypertension in adults. Am Fam Physician. 2014 Oct 1;90(7):503-4. No abstract available. PMID 25369633